CLINICAL TRIAL: NCT01772095
Title: A 6 Months, Prospective, Open-label, Observational, Non-interventional Clinical Trial to Examine the Efficacy and Safety of Donepezil (Dementis®) Administration in Patients With Dementia.
Brief Title: ADVANCE Study: Alzheimer Disease eVAluation iN Clinical PracticE
Acronym: ADVANCE
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-DON-EL-33
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer Disease; Dementia; Cognitive Disorders
Keywords: Donepezil (Dementis); Elderly
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Dementia: Patients diagnosed with dementia and evaluated by specific Alzheimer disease scales

SUMMARY:
In 1906, Dr. Alois Alzheimer first described the disease that later took his name. Today, 100 years later, 24 million people worldwide suffer from Alzheimer's disease or other dementias.

The term 'dementia' is clinical and is used to describe brain disorders that cause decline in mental functions, memory first and then speech, judging and overall behavior. Alzheimer's disease is by far the most common form of dementia, followed by vascular dementia, dementia with Lewy, the frontotemporal dementias etc.

In Greece there are 141,000 patients with dementia. With increasing life expectancy, the figures are expected to increase dramatically in the future.

Alzheimer's disease is the most common form of dementia, as well as 50-60% of patients with dementia suffer from this disease. The second most common type of dementia is vascular, ie that associated with cerebrovascular disease and is the 15-30% of all dementia cases and is most common between the ages of 60-70 years and is more common in men than women. It is estimated that 5% to 8% of people over 65 suffer from dementia, while in industrialized countries ranges at the following levels :15-25% over 85 and 32% over 90 years.

Dementia is characterized by a slow onset and progressive course. The syndrome includes disorders in general intelligence, learning and memory, problem solving, perception, judgment, executive function, language and synergy of movement, but without impairment of consciousness.

Alzheimer's disease is a neurodegenerative disorder with distinct clinical and histopathological features, although with variations from person to person.

In its early stages it is sometimes difficult to diagnose cognitive impairment from normal aging of the brain. With the passage of time, the continuous decline in recent memory, fluency, ability for spatial orientation ultimately restricts the autonomy regarding basic activities of daily life such as managing finances. The anxiety and depression complicate diagnosis in early stages, but gradually decline with loss of sensitivity. Intermediate stages of the disease require increasingly supervision in daily self-care activities, such as personal hygiene and clothing. In the advanced stages are usually essential nursing care in institutional context.

The severity of symptoms of the disease varies and is determined by premorbid factors such as education, gender, cultural background. Epidemiological studies have shown as protective factors against the onset of dementia, higher education, taking estrogen and anti-inflammatory drugs. On the other hand, age, family history of dementia, head injury, hypertension and Down syndrome are risk factors for developing the disease. Finally, some genetic factors appear to be protective, and other pressures to the disease.

DETAILED DESCRIPTION:
Current treatments aim to control the symptoms of the disease. Important parameter is the early diagnosis and early care. The delay in onset of symptoms five years would reduce the incidence of disease by 50% per generation, while complementary therapies and delay entry into institutions would reduce costs considerably. This is the rationale of medication, currently until it causative treatment. The cost of dementia to society as intolerable by the year 2030 it is estimated that a 20% of the population will be over 65. Thus e.g. cost of $ 15 billion currently available in the U.S. for the care of people with dementia are likely to rise further.

Challenge of tackling Alzheimer disease is slowing the degenerative disease process, influencing with any pharmaceutical interventions in various parameters involved in the degeneration of the neuron, resulting in no further for a short-time-charge of the patient's cognition and - the possible load-relief of the family.

Cholinesterase inhibitors are now a documented, effective treatment of the symptoms of Alzheimer disease and therefore are appropriate pharmaceutical intervention. Donepezil has been shown to help and behavioral problems of dementia.

Aging and Dementia Aging as a biological phenomenon leads to irreversible morphologic changes in all body systems. The changes are related to the nervous system can eventually lead to dementia. The population of elderly people is increasing in all developed countries, thereby creating a variety of social, economic and mainly medical problems. This finding has brought interest has to those pathological conditions which are manifested by symptoms that have some qualitative similarity to those of old age and thus both contribute to further expansion in the number of this group of the population and also create diagnostic problems. Morphological, neurochemical and neuropsychological changes that occur in normal aging and dementia observed, especially in Alzheimer.

Dementias are costly illnesses. In Europe today, the cost of care for people with dementia exceeds the cost of illnesses such as heart disease, cancer and strokes.

The last 20 years have been tremendous advances in the prevention, diagnosis and treatment of dementia.

Have significantly increased our knowledge of the predisposing factors of the disease, which helps to prevent. The control of vascular risk factors (hypertension, obesity, diabetes mellitus, hypercholesterolemia, smoking) is beneficial for both the brain and the cardiovascular system. Diet low in fat, fish and vegetarian consumption associated with decreased risk of Disease Alzheimer.

The diagnosis at early clinical stages is possible. An experienced physician can diagnose Alzheimer's with certainty up to 90% by combining the diagnostic tools at his disposal (neuroimaging methods, biomarkers, genetic testing). The pathological process in the brain of patients with Alzheimer's disease begins decades before the appearance of clinical symptoms. The etiology is probably multifactorial. Today intensively sought ways identification of candidate patients and investigated the possibility of non-specific factors (such as hormones, antioxidant vitamins, or anti-inflammatory agents) can reverse or delay the pathogenic process.

Intercultural, people less educated the incidence of dementia is greater. Specially-designed studies have shown that continuing education in adulthood increases cognitive reserve and probably protects against dementia. Those who exercised spiritually (studying, reading) suffer Alzheimer's disease less frequently or in a milder form. Physical exercise and fitness also contribute significantly to the prevention of dementia.

Today's symptomatic treatment of Alzheimer disease . Our experience with drugs called angiotensin cholinesterases (ARICEPT, EXELON, REMINYL) as with the NMDA antagonist (EBIXA) demonstrated that early initiation of treatment significantly slows disease progression Alzheimer, and other dementia syndromes (Vascular and mixed dementia, dementia with Lewy bodies and Alzheimer's Dementia Parkinson).

There is also the non-drug approach the patient exercises involving memory and attention, cognitive empowerment programs, therapy memories orientation to reality. Knowledge empowerment programs aimed at the exploitation of the cognitive functions of patients who remain at a satisfactory level. By using a wide variety of stimuli and specialized methods appropriately stimulated brain of patients and achieve the desired result.

The dementia in the early stages is not easy to diagnose because the public confuses the symptoms to those of normal aging. Still prevalent misconception that nothing can help these patients.

Recent studies have shown that demented patients are usually examined by a specialist 3 years after experiencing the first symptoms of the disease. This delay in diagnosis and treatment has a negative impact on the progress of the disease. Accurate and early diagnosis of dementia, ensure early intervention, smoother transition stages of the disease and a better quality of life for patients and their families for a longer period of time. It also allows further targeted prevention and treatment strategies, medical or otherwise.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older
* Diagnosis of dementia
* Rating 15<MMSE<24
* The patient has reliable caregivers
* Signed consent form to participate in the study after informed by reliable caregivers of the patient or another witness
* The patient is on treatment with donepezil for at least one month prior to joining the clinical trial

Exclusion Criteria:

* Severe gastrointestinal, kidney, hepatic, endocrine, pulmonary, or hematologic disease.
* Other primary psychiatric or neurological disorder.
* Clinically significant laboratory and ECG abnormalities.
* Participation in another clinical study than this
* Refusal to sign the consent form to participate in the study after informed by reliable caregivers of the patient or another witness
* The patient is on treatment with donepezil for less than a month before its integration in the clinical study

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dementia
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in Alzheimer Disease Evaluation Scales (MMSE, Clock test, IADL)from baseline until the end of the study | -1, 0, 3 months, 6 months
  Efficacy of Donepezil (Dementis) treatment MMSE - MiniMental Scale Examination will be performed to all patients for dementia's stage assessment. The mini-mental state examination (MMSE) is a brief 30-point questionnaire test that is used to screen for cognitive impairment. It is commonly used in medicine to screen for dementia. It is also used to estimate the severity of cognitive impairment and to follow the course of cognitive changes in an individual over time, thus making it an effective way to document an individual's response to treatment.
  Clock Drawing Test will be performed to all patients during study visits. IADL (Instrumental Activities of Daily Life Living) scale will be used during all study visits.

SECONDARY OUTCOMES:
Number of Adverse Events occured during study duration | 0, 3 months, 6 months
  Reporting of adverse events during the study period. Safety of Donepezil (Dementis) treatment MMSE - MiniMental Scale Examination will be performed to all patients for dementia's stage assessment. The mini-mental state examination (MMSE) is a brief 30-point questionnaire test that is used to screen for cognitive impairment. It is commonly used in medicine to screen for dementia. It is also used to estimate the severity of cognitive impairment and to follow the course of cognitive changes in an individual over time, thus making it an effective way to document an individual's response to treatment.
  Clock Drawing Test will be performed to all patients during study visits. IADL (Instrumental Activities of Daily Life Living) scale will be used during all study visits.

OTHER OUTCOMES:
Number of days which the patient has not taken his/her study medication | 0,3,6 months
  Compliance to study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Sakka, MD, Study Director — Hygeia Hospital, Athens, Greece; Vasilios Vagenas, MD, Study Director — Sismanogleio Hospital, Athens, Greece; Konstantinos Vadikollias, MD, Study Director — University hospital of Alexandroupolis, Greece; Konstantina Giannopoulou, MD, Study Director — Laiko Hospital of Athens, Greece; Ioannis Metallinos, MD, Study Director — Patras, Greece; Antonios Mougias, MD, Study Director — Athens, Greece; Ioannis Papatriantaphyllou, MD, Study Director — Athens, Greece; Andreas Tzimos, MD, Study Director — Psychiatry Hospital of Thessaloniki, Greece; Xenophon Fitsoris, MD, Study Director — Papageorgiou hospital of Thessaloniki, Greece; Antonis Politis, MD, Associate Professor, Study Chair — Aiginition University Hospital of Athens; Sokratis G Papageorgiou, MD, Associate Professor, Study Director — Attikon Hospital; Evgenia Katirtzoglou, MD, Principal Investigator — Aiginition University Hospital of Athens; Nikolaos Andronas, MD, Principal Investigator — Attikon University Hospital of Athens; Eleni Margioti, Psychologist, PhD, Principal Investigator — Hygeia Hospital of Athens
Locations (1):
- Aiginition University Hospital, Athens, Greece

REFERENCES:
- [Background] Lopez-Pousa S, Bermejo-Pareja F, Frank A, Hernandez F, Leon T, Rejas-Gutierrez J; ECO. [The effect of donepezil in comparison with conventional treatment on cognitive functioning and the performance of the patient in a prospective cohort of patients with Alzheimer's disease treated in routine clinical practice in Spain]. Rev Neurol. 2010 Nov 16;51(10):577-88. Spanish. PMID 21069636
- [Background] Boada-Rovira M, Brodaty H, Cras P, Baloyannis S, Emre M, Zhang R, Bahra R; 322 Study Group. Efficacy and safety of donepezil in patients with Alzheimer's disease: results of a global, multinational, clinical experience study. Drugs Aging. 2004;21(1):43-53. doi: 10.2165/00002512-200421010-00004. PMID 14715043
- [Background] Doody RS, Corey-Bloom J, Zhang R, Li H, Ieni J, Schindler R. Safety and tolerability of donepezil at doses up to 20 mg/day: results from a pilot study in patients with Alzheimer's disease. Drugs Aging. 2008;25(2):163-74. doi: 10.2165/00002512-200825020-00008. PMID 18257603
- [Background] Malouf R, Birks J. Donepezil for vascular cognitive impairment. Cochrane Database Syst Rev. 2004;2004(1):CD004395. doi: 10.1002/14651858.CD004395.pub2. PMID 14974068
- [Background] Johannsen P, Salmon E, Hampel H, Xu Y, Richardson S, Qvitzau S, Schindler R; AWARE Study Group. Assessing therapeutic efficacy in a progressive disease: a study of donepezil in Alzheimer's disease. CNS Drugs. 2006;20(4):311-25. doi: 10.2165/00023210-200620040-00005. PMID 16599649
- [Background] Black SE, Doody R, Li H, McRae T, Jambor KM, Xu Y, Sun Y, Perdomo CA, Richardson S. Donepezil preserves cognition and global function in patients with severe Alzheimer disease. Neurology. 2007 Jul 31;69(5):459-69. doi: 10.1212/01.wnl.0000266627.96040.5a. PMID 17664405
- [Background] Birks J, Harvey RJ. Donepezil for dementia due to Alzheimer's disease. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD001190. doi: 10.1002/14651858.CD001190.pub2. PMID 16437430
- [Background] Matthews HP, Korbey J, Wilkinson DG, Rowden J. Donepezil in Alzheimer's disease: eighteen month results from Southampton Memory Clinic. Int J Geriatr Psychiatry. 2000 Aug;15(8):713-20. doi: 10.1002/1099-1166(200008)15:83.0.co;2-i. PMID 10960883
- [Background] Gauthier S, Feldman H, Hecker J, Vellas B, Ames D, Subbiah P, Whalen E, Emir B; Donepezil MSAD Study Investigators Group. Efficacy of donepezil on behavioral symptoms in patients with moderate to severe Alzheimer's disease. Int Psychogeriatr. 2002 Dec;14(4):389-404. doi: 10.1017/s104161020200858x. PMID 12670060
- [Background] Tricco AC, Vandervaart S, Soobiah C, Lillie E, Perrier L, Chen MH, Hemmelgarn B, Majumdar SR, Straus SE. Efficacy of cognitive enhancers for Alzheimer's disease: protocol for a systematic review and network meta-analysis. Syst Rev. 2012 Jun 28;1:31. doi: 10.1186/2046-4053-1-31. PMID 22742585
- [Background] Tariot P, Salloway S, Yardley J, Mackell J, Moline M. Long-term safety and tolerability of donepezil 23 mg in patients with moderate to severe Alzheimer's disease. BMC Res Notes. 2012 Jun 8;5:283. doi: 10.1186/1756-0500-5-283. PMID 22681723
- [Background] Isik AT, Yildiz GB, Bozoglu E, Yay A, Aydemir E. Cardiac safety of donepezil in elderly patients with Alzheimer disease. Intern Med. 2012;51(6):575-8. doi: 10.2169/internalmedicine.51.6671. Epub 2012 Mar 15. PMID 22449664
- [Background] Rungsanpanya T, Muangpaisan W, Praditsuwan R. Clinical practice with antidementia drugs in a geriatric clinic. J Med Assoc Thai. 2012 Aug;95(8):1081-9. PMID 23061314
- [Background] Isik AT, Bozoglu E, Yay A, Soysal P, Ateskan U. Which cholinesterase inhibitor is the safest for the heart in elderly patients with Alzheimer's disease? Am J Alzheimers Dis Other Demen. 2012 May;27(3):171-4. doi: 10.1177/1533317512442999. PMID 22573283
- [Background] Bond M, Rogers G, Peters J, Anderson R, Hoyle M, Miners A, Moxham T, Davis S, Thokala P, Wailoo A, Jeffreys M, Hyde C. The effectiveness and cost-effectiveness of donepezil, galantamine, rivastigmine and memantine for the treatment of Alzheimer's disease (review of Technology Appraisal No. 111): a systematic review and economic model. Health Technol Assess. 2012;16(21):1-470. doi: 10.3310/hta16210. PMID 22541366